CLINICAL TRIAL: NCT01230866
Title: A Phase III Prospective Randomized Trial of Standard-fractionation vs. Hypo-fractionation With Proton Radiation Therapy for Low Risk Adenocarcinoma of the Prostate
Brief Title: Study of Hypo-fractionated Proton Radiation for Low Risk Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Proton Collaborative Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GU002-10
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Proton Radiation Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proton Radiation Hypofractionation (Other): 5 fractions (7.6 Gy(RBE) x 5)
  Interventions: Radiation: Proton Radiation Hypofractionation
- Proton Radiation Standard Fractionation (Active Comparator): 44 fractions (1.8 Gy(RBE) x 44)
  Interventions: Radiation: Proton Radiation Standard Fractionation

INTERVENTIONS:
Radiation: Proton Radiation Hypofractionation — Dose: 38 Gy(RBE); 7.6 GY(RBE) five days a week in 5 treatments over 1-2 weeks
  Other Names: Particle Therapy
  Arms: Proton Radiation Hypofractionation
Radiation: Proton Radiation Standard Fractionation — Dose: 79.2 GY(RBE); 1.8 GY(RBE) five days a week in 44 treatments over 8.5-9 weeks
  Other Names: Particle Therapy
  Arms: Proton Radiation Standard Fractionation

SUMMARY:
The purpose of this study is to compare the effects (good and bad) on patients with prostate cancer by comparing the standard dose of radiation therapy (44 treatments over 8½-9 weeks) with a higher daily dose of radiation (5 treatments over 1-2 weeks) to see if the effects of the treatments are similar or better.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma within 365 days prior to randomization.
* History/physical examination with digital rectal examination of the prostate and baseline toxicity assessment within 90 days prior to randomization.
* Histological evaluation of prostate biopsy with assignment of a Gleason score to the biopsy material;Gleason score must be in the range of 2-6. > 6 cores are strongly recommended.
* PSA values < 10 ng/ml within 90 days prior to randomization. Either done prior to biopsy or at least 21 days after prostate biopsy.
* Clinical stages T1a-T2a N0 M0 (AJCC Criteria 7th Ed.). Staging must be done by treating investigator.
* No pelvic lymph nodes > 1.5 cm in greatest dimension unless the enlarged lymph node is biopsied and negative.
* Patients must be at least 18 years old.
* ECOG performance status 0-1 (appendix I) documented within 90 days prior to randomization.
* IPSS score <= 16.
* Patients must give IRB approved, study specific, informed consent.
* Patients must complete all mandatory tests listed in section 4.0 within the specified time frames.
* Patients must be able to start treatment within 56 days of randomization.

Exclusion Criteria:

* Previous prostate cancer surgery to include: prostatectomy, hyperthermia and cryosurgery.
* Previous pelvic radiation for prostate cancer.
* Androgen deprivation therapy prior to radiation is allowed. However, it is not acceptable if continued during radiation or as adjuvant therapy.
* Active rectal diverticulitis, Crohn's disease affecting the rectum, or ulcerative colitis.
* Prior systemic chemotherapy for prostate cancer.
* History of proximal urethral stricture requiring dilatation.
* Current and continuing anticoagulation with warfarin sodium (Coumadin, heparin, low-molecular weight heparin, Clopidogrel bisulfate (Plavix),or equivalent. (Unless it can be stopped to manage treatment related toxicity, to have a biopsy if needed, or for marker placement).
* Any major medical, addictive or psychiatric illnesses which would affect the consent process, completion of treatment and/or interfere with follow-up. Consent by legal authorized representative is not permitted in this study.
* Evidence of any other cancer within the past 5 years and < 50% probability of a 5 year survival. (Prior or concurrent diagnosis of basal cell or non-invasive squamous cell cancer of the skin is allowed).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-11; Primary Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To assess if hypo-fractionation will result in 2-year freedom from failure (FFF) that is non-inferior to 2-year FFF following standard fractionation. FFF will be measured by recurrence, metastasis, PSA or start of salvage therapy. | At 5 years post treatment completion +/- 90 days
  The events for FFF will be the first occurrence of clinical failure (local recurrence, regional recurrence, or distant metastasis), biochemical failure by the Phoenix definition (PSA ≥ 2 ng/ml over the current nadir PSA),or the start of salvage therapy including androgen deprivation.

SECONDARY OUTCOMES:
To determine the incidence of grade 2 or greater GU and GI toxicity in each of the regimens. | At 6 months and 2 years post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Vargas, MD, Study Chair — Proton Collaborative Group
Locations (5):
- United States (5):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - Northwestern Medicine Chicago Proton Center, Warrenville, Illinois
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - Oklahoma Proton Center, Oklahoma City, Oklahoma
  - Hampton University Proton Therapy Institute, Hampton, Virginia

REFERENCES:
- [Derived] Toesca DAS, Hartsell WF, DeWees TA, Chang JH, Laughlin BS, Voss MM, Dodoo CA, Mohammed N, Keole SR, McGee LA, Gondi V, Sweeney PJ, Dorn P, Sinesi CC, Doh LS, Rich T, Vargas CE. Stereotactic Body Proton Therapy Versus Conventionally Fractionated Proton Therapy for Early Prostate Cancer: A Randomized, Controlled, Phase 3 Trial. Int J Radiat Oncol Biol Phys. 2024 Dec 1;120(5):1377-1385. doi: 10.1016/j.ijrobp.2024.05.014. Epub 2024 Jul 6. PMID 38972465